CLINICAL TRIAL: NCT07051941
Title: Validation of a User Questionnaire to Assess Surgeon Satisfaction and Perspectives on Robotic Surgical Systems (Robotic Surgeon Satisfaction Questionnaire - RSSQ)
Brief Title: Validation of a User Questionnaire to Assess Surgeon Satisfaction and Perspectives on Robotic Surgical Systems
Acronym: RSSQ
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 7809
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Surgery
Keywords: robotic surgery; robotic system; precision; ergonomics; safety

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgeon: The validation study will include a cohort of expert robotic surgeons (n = ~50-100) who have performed at least 100 robotic procedures with one or more platforms (Da Vinci®, Hugo™, etc.). Inclusion criteria:
  * Board-certified surgeons
  * At least 1 year of experience with robotic-assisted surgery
  * Informed consent to participate
  Interventions: Other: Validation of a satisfaction questionnaire for robotic surgeon

INTERVENTIONS:
Other: Validation of a satisfaction questionnaire for robotic surgeon — The primary endpoint is to validate a questionnaire to assess user satisfaction among expert surgeons utilizing various surgical robotic systems, including - but not limited to - the Da Vinci®, Hugo™ RAS, Versius®, and Toumai® platforms.
  Based on these domains, an initial pool of items was generated; items were formulated as Likert-scale questions (5-point) and grouped into thematic sections.
  The validation of the Questionnaire will be developed with a 2-step process.
  1. Test for Content Validity and Face Validity: a pilot test will be performed with 5-10 surgeons from FPG to ensure content and face validity, item comprehension, and usability.
  2. Validation from external users:

SUMMARY:
Robotic surgery represents a cornerstone for surgical treatment of different diseases. Since the Da Vinci patent expiry, several new robotic systems entered the market in the effort to spread to a greater extent the benefits of robotic surgery. Even if clinical comparison between new systems and the Da Vinci platform are currently available, there is lack of reporting about subjective perception of surgeons approaching new platforms; personal feedback on fluency and precision, ergonomics, OR communication and other items are missing.The aim of the study is to validate a practical, reproducible, and comparable instrument that can be applied in both clinical research and in the evaluation processes of newly introduced surgical robotic platforms.

DETAILED DESCRIPTION:
In recent years, the expansion of the robotic surgery landscape has been marked by the introduction of several new systems alongside the well-established Da Vinci platform. Emerging technologies such as Hugo™, Versius™, and Toumai™ offer distinct features in terms of ergonomics, system flexibility, user interface, and integration within the intraoperative workflow.

Initial comparison between new systems and the Da Vinci platform are currently available and include both clinical [1] and cost comparison [2,3]. However, there is a lack of reporting about subjective perception of surgeons approaching new platforms; personal feedback on fluency and precision, ergonomics, OR communication and other items are missing.

Some studies tried to address the issue [4-7]; however, to now, no instrument able to evaluate users' satisfaction on different robotic system is available.

Thus, there is a growing need for standardized tools capable of capturing the surgeon's subjective experience when using a specific robotic platform.

The present study aims to develop and validate a user satisfaction questionnaire for surgeons who operate with robotic systems, with the goal of assessing both qualitative and quantitative aspects related to perceived reliability and safety, movement fluency, ergonomic comfort, communication with staff, ease of setup (docking), and overall satisfaction.

In this evolving landscape, standardized tools are essential to assess surgeons' subjective perceptions regarding the use of specific robotic platforms. User satisfaction is a critical indicator for the adoption and effectiveness of new surgical technologies.

The aim of the study is to provide a practical, reproducible, and comparable instrument that can be applied in both clinical research and in the evaluation processes of newly introduced surgical robotic platforms.

STUDY OBJECTIVE

This study aims to validate a surgeon satisfaction questionnaire for those surgeons utilizing robotic surgical systems. The goal is to evaluate qualitative and quantitative aspects related to:

* Perceived reliability and safety
* Movement fluidity
* Ergonomics and physical comfort
* Communication with staff
* Ease of setup (docking)
* Overall satisfaction The questionnaire has been developed by two surgeons (MCS and BR) for the evaluation of a single robotic system and could be intended as "procedure-specific" or it could also be used to assess the overall and comprehensive performance of the platform (non-procedure specific).

The questionnaire does not represent itself a tool for the comparison of new robotic systems; however, its outcome measures are objective and could be used for the comparative evaluation of robotic systems. The questionnaire could be applied to surgeons of different disciplines (urology; general surgery; gynecology; etc).

METHODS Study Design This study follows a cross-sectional design. The primary endpoint is to validate a questionnaire to assess user satisfaction among expert surgeons utilizing various surgical robotic systems, including - but not limited to - the Da Vinci®, Hugo™ RAS, Versius®, and Toumai® platforms.

The Questionnaire has been developed from two Authors (MCS and BR) according to the following steps:

1. Literature Review and Domain Identification

   A comprehensive literature review was conducted to identify key domains related to user satisfaction with robotic surgical systems. Major areas identified include:
   * System reliability and precision
   * Ease of setup and docking
   * Instrument and console ergonomics
   * System-team communication
   * Intuitive control and usability
   * Visual quality and haptics
   * Workflow fluency
   * Perceived safety and trust in technology
2. Item Generation Based on these domains, an initial pool of items was generated; items were formulated as Likert-scale questions (5-point) and grouped into thematic sections. Both positive and negative phrasing was used to reduce response bias. An draft of the survey is reported as Supplementary Material.

The validation of the Questionnaire will be developed with a 2-step process.

1. Test for Content Validity and Face Validity: a pilot test will be performed with 5-10 surgeons from FPG to ensure content and face validity, item comprehension, and usability.
2. Validation from external users:

Participants

The validation study will include a cohort of expert robotic surgeons (n = ~50-100) who have performed at least 100 robotic procedures with one or more platforms (Da Vinci®, Hugo™, etc.). Inclusion criteria:

* Board-certified surgeons
* At least 1 year of experience with robotic-assisted surgery
* Informed consent to participate Participants will be recruited on a voluntary basis from the boards/members of international scientific societies (ERUS Scientific Working Group - European Robotic Urology Section; Agile Group; Society of Robotic Surgery); surgeons will be enrolled from high-volume surgical centers in Europe, North America, and Asia, South America, Africa.

Data Collection Surgeons will be invited to complete the questionnaire via a secure web-based platform (Survey Monkey). The on-line questionnaire will start with a brief explanation of the project and with the Informed Consent to be signed from the surgeon to participate in the study; if denied, the questionnaire will be automatically deleted. If the surgeon agrees to participates, the questionnaire will develop according to the attached Supplementary File. Demographic data (age, gender, years of robotic experience, surgical specialty, platform used) will also be collected.

Statistical analysis Reliability Analysis

* Internal consistency will be assessed using Cronbach's alpha for each domain. A threshold of α ≥ 0.70 will be considered acceptable.
* Item-total correlations and inter-item correlations will be examined. Construct Validity
* Exploratory Factor Analysis will be performed using principal component analysis with varimax rotation to identify the latent structure of the questionnaire.
* The Kaiser-Meyer-Olkin measure and Bartlett's test of sphericity will assess data suitability for factor analysis.

Test-Retest Reliability A subgroup of surgeons (n = 20) will be asked to complete the questionnaire twice, 1-2 weeks apart. Intraclass Correlation Coefficient (ICC) will be calculated to evaluate temporal stability.

ELIGIBILITY:
Inclusion Criteria:

* Board-certified surgeons
* At least 1 year of experience with robotic-assisted surgery
* Signed informed consent to participate

Exclusion Criteria:

* Participants not fitting inclusion criteria
* Unwilling to participate

Ages: 30 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participant surgeons will be recruited among scientific organization/communities focused on robotic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Internal consistency. | 6 months
  Internal consistency: assessed using Cronbach's alpha for each domain. A threshold of α ≥ 0.70 will be considered acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Maria chiara Sighinolfi, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS

IPD SHARING:
Plan to Share IPD: Undecided